CLINICAL TRIAL: NCT02556502
Title: 18F-Florbetaben PET Amyloid Imaging in Case of Intermediate CSF Biology for the Diagnosis of Alzheimer's Disease : a Pilot Study
Acronym: MAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-A01149-40
Record Dates: First submitted 2015-09-21; First posted 2015-09-22 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Amyloid PET Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FDG PET positive or negative (Experimental)
  Interventions: Device: 18F-Florbetaben PET

INTERVENTIONS:
Device: 18F-Florbetaben PET

SUMMARY:
The diagnosis of Alzheimer's disease (AD) is based on clinical and neuropathological criteria.

Some patients have a contributive CSF biology to determinate a high level risk of AD (Tau + phospho-tau ratio increased and Ab42 / decreased Aβ40), but others have an intermediate CSF biology (Tau and/or phospho-tau increased but Ab42 ratio / normal Aβ40) and are unclassifiable.

18F-Florbetaben (Neuraceq®), a radioisotope in positron emission tomography (PET), selectively binds to amyloid plaques, with high detection sensitivity (98%).

Detection of amyloid plaques by PET imaging separate patients according to the criteria of Dubois, as with AD and allow them to benefit a cholinesterase inhibitor treatment.

If negative, the diagnosis of AD can be excluded with a high level of confidence to prevent initiating unnecessary treatment, expensive for the community.

This is the first imaging study of amyloid plaques targeting population whose diagnosis of AD is uncertain according to the CSF biology.

The aim of this study is to describe the results of amyloid PET in case of intermediate CSF biology and to separate patients as AD or not according to the criteria of Dubois

ELIGIBILITY:
Inclusion Criteria:

* Major subjects who have given their consent to participate in the study.
* Patients with suspected AD and whose CSF markers give intermediate results (CSF punction less than 6 months): meaning tau and/or phospho-tau increased and Ab42 / Aβ40 normal (Ab42 / Aβ40 > 0.07).
* Non-indication to perform a PET 18F-Florbetaben.
* Affiliation to the french social security .

Exclusion Criteria:

* Patients under guardianship.
* Inability to perform a PET 18F-Florbetaben (agitated patient, confused, ..).
* Pregnancy, lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-11; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
number of positive or negative amyloid PET | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Vandœuvre-lès-Nancy, France